CLINICAL TRIAL: NCT05385211
Title: CFTR and Exocrine Pancreatic Dysfunction in Type 1 Diabetes
Brief Title: Cystic Fibrosis Transmembrane Conductance Regulator (CFTR) and Exocrine Pancreatic Dysfunction in Type 1 Diabetes
Status: Completed | Type: Observational
Sponsor: Ciusss de L'Est de l'Île de Montréal (Other)
Collaborators: Juvenile Diabetes Research Foundation (Other); Institut de Recherches Cliniques de Montreal (Other)
Responsible Party: Principal Investigator, Sylvie Lesage, Principal investigator, Ciusss de L'Est de l'Île de Montréal
Other Study IDs: 1-INO-2022-1126-A-N
Record Dates: First submitted 2022-05-17; First posted 2022-05-23 (Actual); Last update posted 2023-09-05 (Actual); Status verified 2023-09

CONDITIONS: Type 1 Diabetes; Exocrine Pancreatic Insufficiency
Keywords: Cystic fibrosis transmembrane regulator; Type 1 diabetes; Hypoglycemia; Exocrine pancreas
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Exocrine Pancreatic Insufficiency; Hypoglycemia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Blood sampling
  Data from continuous glucose monitoring
  DNA for CFTR sequencing
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- People living with type 1 diabetes: Participants will be separated into two groups based on the levels of their exocrine pancreatic enzymes levels.
  Interventions: Other: Frequency of hypoglycemia in people with type 1 diabetes and exocrine pancreatic insufficiency

INTERVENTIONS:
Other: Frequency of hypoglycemia in people with type 1 diabetes and exocrine pancreatic insufficiency — Blood samplings; Glucose monitoring; CFTR variants

SUMMARY:
This study proposes to examine the contribution of CFTR variants to exocrine pancreatic insufficiency and hypoglycemic risk. Hypoglycemia is one the most frequent complications of type 1 diabetes management. Despite recent innovations, hypoglycemic risk remains high for people living with type 1 diabetes (PWT1D). Recent studies have shown that pancreatic insufficiency could affect hypoglycemic risk. Up to now, there are limited data on the association between pancreatic insufficiency and glucose control (i.e. the frequency and severity of hypoglycemic episodes as well as HbA1c levels). The main objective of this study is to determine the impact of pancreatic insufficiency on glucose control in PWT1D, and to address the role of CFTR variants as potential contributors to pancreatic insufficiency.

DETAILED DESCRIPTION:
In this a one year cross sectional study, we plan to enroll 100 adults living with type 1 diabetes.

Patient data will then be separated into two groups based the presence or absence of exocrine pancreatic insufficiency (EPI). EPI will be defined based on the levels of pancreatic enzymes (Amylase; lipase; and trypsinogen). As the prevalence of EPI in people living with type 1 diabetes (PWT1D) is ~50%, we expect roughly the same number of individuals into both groups (with or without EPI).

Variables :

Subject data (age, gender, duration of diabetes, age at diagnostic, etc.) will be collected.

Glucose variation will be assessed with a continuous glucose monitoring system for 1 month. Briefly we will collect the number and severity of hyperglycemic events, average glucose levels, glycemic variability, etc..

From collected peripheral blood mononuclear cells (PBMCs) we will quantify CFTR function and level of expression, as well as identify CFTR variants by next generation sequencing.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 diabetes
* Living in Montreal

Exclusion Criteria:

* Pregnancy,
* Use of corticosteroid
* Use of medication known to have a relevant impact on glycemic control.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: People living with type 1 diabetes
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2022-04-30 (Actual); Primary Completion 2023-08-30 (Actual); Study Completion 2023-08-30 (Actual)

PRIMARY OUTCOMES:
Frequency and severity of hypoglycemic events | 1 month
  Continuous glucose monitoring will be used to assess glucose regulation
Exocrine pancreatic insufficiency | Baseline
  Blood levels of pancreatic enzymes will be measured

CONTACTS AND LOCATIONS:
Overall Officials: Sylvie Lesage, Ph.D, Principal Investigator — Ciusss de L'Est de l'Île de Montréal
Locations (1):
- Institut de recherches cliniques de Montréal, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No